CLINICAL TRIAL: NCT02420314
Title: A Phase II Trial of High-Dose Ascorbate in Stage IV Non-Small Cell Lung Cancer
Brief Title: Pharmacological Ascorbate for Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph J. Cullen, MD, FACS (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); Holden Comprehensive Cancer Center (Other); McGuff Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Muhammad Furqan, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201412760; 3P30CA086862 (NIH)
Record Dates: First submitted 2015-04-09; First posted 2015-04-17 (Estimated); Results first posted 2024-04-17 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Ascorbate; Ascorbic acid; Vitamin C; NSCLC; Non Small Cell Lung Cancer; carboplatin; paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Carboplatin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ascorbate, paclitaxel, carboplatin (Experimental): Paclitaxel, administered once per cycle (3 weeks) Carboplatin, administered once per cycle (3 weeks) Pharmacological ascorbate (ascorbic acid) infusions, 2 times per week for 3 weeks
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Paclitaxel — * Administered intravenously (IV)
  * Prescribed at 200 mg/m2 (standard dose)
  * Given once every 21 days (i.e., one cycle)
  * Up to 4 cycles are administered depending on disease response
  Other Names: Nov-Onxol; Onxol; Paclitaxel Novaplus; Taxol
Drug: Carboplatin — * Administered intravenously (IV)
  * Prescribed at AUC = 6 using the Cockcroft-Gault formula (standard dose)
  * Given once every 21 days (i.e., one cycle)
  * Up to 4 cycles are administered depending on disease response
  Other Names: Amerinet Choice Carboplatin; NovaPlus CARBOplatin; Paraplatin; Paraplatin NovaPlus
Drug: Ascorbic Acid — * Administered intravenously (IV)
  * 75g per infusion
  * Two infusions per week
  * 1 cycle is 3 weeks
  * given up to 4 cycles
  * may be given while chemotherapy if delayed due to low counts
  Other Names: Pharmacological ascorbate; Vitamin C; Ascorbate

SUMMARY:
This clinical trial evaluates adding high-dose ascorbate (vitamin C) to standard of care treatment of non-small cell lung cancer (NSCLC) in adults. All subjects will receive high-dose ascorbate in addition to the standard treatment.

DETAILED DESCRIPTION:
Standard treatment for non-small cell lung cancer (NSCLC) involves a combined therapy of paclitaxel and carboplatin. These drugs are administered once every 21 days. This study adds high dose ascorbic acid (75g per infusion) twice per week for up to 4 cycles of therapy.

Participants will:

* receive high doses of intravenous (IV) ascorbate two times a week during each 3 week chemotherapy.
* have blood samples drawn to measure blood ascorbate levels once every 21 days
* have blood samples drawn to measure iron and ferritin levels before treatment, then on cycles 1 and 3.

The active therapy portion of this study lasts for 4 months. After that is completed, participants will go back to standard therapy for their cancer. Participants will continue to have life-long follow-up for this study.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed stage IIIB or IV non -small cell lung cancer. The potential participant must not have received first-line cytotoxic therapy. Prior use of first-line EGFR inhibitors or ALK inhibitors is allowed if there was progression on therapy.
* CNS metastasis is allowed if the metastasis is treated and there are no signs of progression following treatment. The potential participant must be off steroids for at least 3 days and be stable.
* At least 18 years of age
* ECOG performance status of 0, 1, or 2
* absolute neutrophil count (ANC) of at least 1500 cells per mm³
* platelet count of at least 100,000 cells per mm³
* hemoglobin of at least 8 g/dL
* creatinine within 1.5 times the upper limit of normal
* total bilirubin within 1.5 times the upper limit of normal
* ALT within 3 times the institutional upper limit of normal
* AST within 3 times the institutional upper limit of normal
* the participant must tolerate a 15g ascorbate test infusion (screening dose)
* patients who received prior treatment with curative intent must have experienced a treatment-free interval of at least 6 months since the last treatment
* the participant must not be pregnant, be willing to have a pregnancy test done if deemed necessary, and be willing to use adequate birth control during the study
* not breastfeeding
* independently able to provide consent (legally authorized representative and/or power of attorney is not allowed)

Exclusion Criteria:

* known sensitizing EGFR mutations or ALK gene rearrangements if the participant has not yet tried EGFR or ALK inhibitor therapies. If the potential participant's biopsy did not allow for gene analysis (inconclusive, not enough tissue), the patient is considered eligible for the study. Enrollment on this clinical trial after progression on targeted therapy is allowed
* 50% or greater PD-L1 expression (patients with unknown PD-L1 expression or when PD-L1 expression can't be determined due to insufficient tumor sample or other reasons remain eligible)
* receiving warfarin therapy and cannot tolerate drug substitution
* active hemoptysis within 1 week of screening (more than 1/2 teaspoon of blood per day)
* actively receiving insulin at the time of ascorbate infusion
* G6PD deficiency
* leptomeningeal disease
* potential participants cannot be on the following drugs: flecainide, methadone, amphetamines, quinidine, or chlorpropamide.
* known active invasive malignancy other than the lung cancer under therapy (non-melanoma skin cancer or carcinoma in situ of the cervix or bladder are exempted)
* potential participants may not enroll in, or be actively receiving treatment from, a therapeutic clinical trial for their cancer. Observational studies (including imaging studies) are acceptable.
* uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness / social situations that would limit compliance with study requirements
* known HIV positive individuals cannot be enrolled in this trial because high-dose ascorbate is a known CYP450 3A4 inducer, which results in lower serum levels of antiretroviral agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Cullen, MD, FACS, Study Director — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared from those patient partners who agree to it. Data will be codified for the investigational team to provided additional details - as necessary - or confirm against source.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: Email the study chair or principal investigator; a non-disclosure and/or data usage agreement will most likely be required.

REFERENCES:
- [Result] Schoenfeld JD, Sibenaller ZA, Mapuskar KA, Wagner BA, Cramer-Morales KL, Furqan M, Sandhu S, Carlisle TL, Smith MC, Abu Hejleh T, Berg DJ, Zhang J, Keech J, Parekh KR, Bhatia S, Monga V, Bodeker KL, Ahmann L, Vollstedt S, Brown H, Shanahan Kauffman EP, Schall ME, Hohl RJ, Clamon GH, Greenlee JD, Howard MA, Schultz MK, Smith BJ, Riley DP, Domann FE, Cullen JJ, Buettner GR, Buatti JM, Spitz DR, Allen BG. O2⋅- and H2O2-Mediated Disruption of Fe Metabolism Causes the Differential Susceptibility of NSCLC and GBM Cancer Cells to Pharmacological Ascorbate. Cancer Cell. 2017 Apr 10;31(4):487-500.e8. doi: 10.1016/j.ccell.2017.02.018. Epub 2017 Mar 30. PMID 28366679
- [Result] Furqan M, Abu-Hejleh T, Stephens LM, Hartwig SM, Mott SL, Pulliam CF, Petronek M, Henrich JB, Fath MA, Houtman JC, Varga SM, Bodeker KL, Bossler AD, Bellizzi AM, Zhang J, Monga V, Mani H, Ivanovic M, Smith BJ, Byrne MM, Zeitler W, Wagner BA, Buettner GR, Cullen JJ, Buatti JM, Spitz DR, Allen BG. Pharmacological ascorbate improves the response to platinum-based chemotherapy in advanced stage non-small cell lung cancer. Redox Biol. 2022 Jul;53:102318. doi: 10.1016/j.redox.2022.102318. Epub 2022 Apr 20. PMID 35525024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was between April 2015 through November 2020
Groups:
- Ascorbate, Paclitaxel, Carboplatin: Paclitaxel, administered once per cycle (3 weeks) Carboplatin, administered once per cycle (3 weeks) Pharmacological ascorbate (ascorbic acid) infusions, 2 times per week for 3 weeks
  Paclitaxel: - Administered intravenously (IV)
  * Prescribed at 200 mg/m2 (standard dose)
  * Given once every 21 days (i.e., one cycle)
  * Up to 4 cycles are administered depending on disease response
  Carboplatin: - Administered intravenously (IV)
  * Prescribed at AUC = 6 using the Cockcroft-Gault formula (standard dose)
  * Given once every 21 days (i.e., one cycle)
  * Up to 4 cycles are administered depending on disease response
  Ascorbic Acid: - Administered intravenously (IV)
  * 75g per infusion
  * Two infusions per week
  * 1 cycle is 3 weeks
  * given up to 4 cycles
  * may be given while chemotherapy if delayed due to low counts
Period: Overall Study
Arm/Group | Ascorbate, Paclitaxel, Carboplatin
Started | 40
Completed | 38
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ascorbate, Paclitaxel, Carboplatin
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — Self-declared gender
  Participants
    Female | 13
    Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported race & ethnicity
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 37
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: From cycle 1, day 1, to documented disease progression in CT imaging as described by RECIST criteria
Time Frame: every 2 months for up to 5 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ascorbate, Paclitaxel, Carboplatin
Number analyzed (Participants) | 38
Participants
  confirmed partial response | 13
  stable disease | 19
  progressive disease | 5
  unevaluable | 1

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The time (in months) it takes for disease to progress as defined by RECIST criteria. Timeframe will be from cycle 1, day 1 to date of progression.
Time Frame: every 2 months for up to 5 years post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ascorbate, Paclitaxel, Carboplatin
Number analyzed (Participants) | 38
months | 5.7 [4.3 to 7.0]

3. Secondary Outcome: Overall Survival (OS)
Description: Time, measured in months, from cycle 1 day 1 until date of death from any cause
Time Frame: every 2 months for up to 5 years post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ascorbate, Paclitaxel, Carboplatin
Number analyzed (Participants) | 38
months | 12.8 [8.7 to 21.7]

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 5 years post-treatment. Adverse events were assessed for up to 6 months post-enrollment (minimum of 21 days after the final ascorbate infusion if early completion).
Description: Adverse events are defined by federal code and consistent with the definitions provided by clinicaltrials.gov
Arm/Group | Ascorbate, Paclitaxel, Carboplatin
All-Cause Mortality (participants affected / at risk) | 31/40
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbate, Paclitaxel, Carboplatin (N=40)
Cardiac disorder, other (Cardiac disorders) | 1 (1) — T-wave inversion
urinary tract infection (Infections and infestations) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
urinary retention (Renal and urinary disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
lung infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Community acquired pneumonia
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
thromboembolic event (Vascular disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
hepatobiliary disorder, other (Hepatobiliary disorders) | 1 (1) — Acute liver injury
Death nos (General disorders) | 1 (1) — probable from renal failure
Fever (General disorders) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ascorbate, Paclitaxel, Carboplatin (N=40)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (7)
Alkaline phosphatase increased (Investigations) | 5 (5)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 23 (23)
Ankle sprain (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 15 (15)
anxiety (Nervous system disorders) | 11 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (16)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
benign prostate hypertrophy (Reproductive system and breast disorders) | 1 (1)
bicarbonate decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
body pain (General disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Burning at IV site (General disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Creatinine increased (Investigations) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Dizziness (Nervous system disorders) | 3 (3)
drowsiness (Nervous system disorders) | 1 (1)
Dry lips (Skin and subcutaneous tissue disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 16 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Ear pain (Ear and labyrinth disorders) | 2 (2)
early satiety (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 4 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
elevated iron (Investigations) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 29 (29)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 8 (8)
Flank pain - right side (Musculoskeletal and connective tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
GGT increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot flash (General disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 15 (15)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (10)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 11 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection - toenail (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 4 (4)
Infusion site extravasation (General disorders) | 1 (1)
Injection site reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Itchy ears (Skin and subcutaneous tissue disorders) | 1 (1)
IV infiltration (General disorders) | 2 (2)
IV site pain (General disorders) | 1 (1)
knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
left big toe pain (Skin and subcutaneous tissue disorders) | 1 (1)
left hip and low back (Musculoskeletal and connective tissue disorders) | 1 (1)
lip bite (Skin and subcutaneous tissue disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 13 (13)
Maculopapular rash (Immune system disorders) | 1 (1)
metatarsal fracture (Injury, poisoning and procedural complications) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
mural thrombus (Vascular disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb right side (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 26 (26)
Neutrophil count decreased (Investigations) | 15 (15)
night sweats (Vascular disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Non-specific T wave abnormality (Cardiac disorders) | 1 (1)
Oral Candidiasis (Infections and infestations) | 2 (2)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 5 (5)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity - bilateral hand (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity - right arm (Musculoskeletal and connective tissue disorders) | 1 (1)
pain left big toe (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
pain over 3 metatarsal LT foot (Musculoskeletal and connective tissue disorders) | 1 (1)
paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1)
Peripheral edema, right arm (General disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 24 (24)
Platelet count decreased (Investigations) | 16 (16)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
port site pain (General disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
RLL pulmonary embolus (Vascular disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Skin infection (Infections and infestations) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 4 (4)
tingling left hand (Nervous system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 13 (13)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 10 (10)

LIMITATIONS AND CAVEATS:
Single arm, open label trial increases bias and reduces internal validity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT02420314/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT02420314/ICF_001.pdf